CLINICAL TRIAL: NCT02822508
Title: A Safety and Efficacy Evaluation of BLI801 Laxative in Adults Experiencing Non-Idiopathic Constipation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BLI801-203
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- BLI801 Laxative (high dose) (Experimental): BLI801 Laxative (high dose)
  Interventions: Drug: BLI801 Laxative
- BLI801 Laxative (mid dose) (Experimental): BLI801 Laxative (mid dose)
  Interventions: Drug: BLI801 Laxative
- BLI801 Laxative (low dose) (Experimental): BLI801 Laxative (low dose)
  Interventions: Drug: BLI801 Laxative
- BLI801 Placebo (Placebo Comparator): BLI801 Placebo
  Interventions: Drug: BLI801 Placebo

INTERVENTIONS:
Drug: BLI801 Laxative — BLI801 oral laxative
  Arms: BLI801 Laxative (high dose); BLI801 Laxative (low dose); BLI801 Laxative (mid dose)
Drug: BLI801 Placebo — BLI801 oral laxative placebo
  Arms: BLI801 Placebo

SUMMARY:
The objective of this study is to evaluate multiple doses of BLI801 Laxative for safety and efficacy versus placebo in adults experiencing non-idiopathic constipation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between the ages of > 18 and < 85 years
2. Constipated, defined by the following criteria: Fewer than 3 spontaneous defecations per week and at least one of the following symptoms for the previous 4 weeks:

   * Straining during > 25% of defecations
   * Lumpy or hard stools in > 25% of defecations
   * Sensation of incomplete evacuation for > 25% of defecations
3. Receiving a stable maintenance opioid regimen.
4. If female, and of child-bearing potential, is using an acceptable form of birth control
5. Negative pregnancy test at screening (Visit 1), if applicable
6. In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study

Exclusion Criteria:

1. Subjects with known or suspected ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis or toxic megacolon
2. Subjects who have had major surgery within 30 days before Visit 1; appendectomy or cholecystectomy 60 days before Visit 1; abdominal, pelvic, or retroperitoneal surgery 6 months before Visit 1; bariatric surgery or surgery to remove a segment of the GI tract at any time before Visit 1
3. Medical conditions associated with diarrhea, intermittent loose stools or constipation, which could confound the interpretation of the results, eg, fecal incontinence or irritable bowel syndrome. Subjects with irritable bowel syndrome (IBS) that has been previously diagnosed by a physician prior to initiation of the constipating therapy and that meets the following criteria, are excluded:

   1. Absence of a structural or biochemical explanation for the abdominal pain symptom
   2. At least 12 weeks during a period of 12 months, of abdominal discomfort or pain with at least 2 of the following 3 features:

   i. Relieved with defecation, and/or ii. Onset associated with a change in frequency of stool, and/or iii. Onset associated with a change in form of stool.
4. Subjects diagnosed with chronic constipation prior to initiation of opioid treatment
5. Subjects taking laxatives (with the exception of fiber supplements), prokinetic agents or antidiarrheal drugs and refuse to discontinue these treatments from Visit 1 until after completion of Visit 5
6. Subjects who are pregnant or nursing, or intend to become pregnant during the study
7. Subjects of childbearing potential who refuse a pregnancy test
8. Subjects who are allergic to any BLI801 component
9. Subjects taking non-opioid medications or supplements known to cause constipation
10. Subjects with an active history of drug or alcohol abuse
11. Subjects who have participated in an investigational clinical, surgical, drug, or device study within the past 30 days
12. Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures.
13. Subjects who have had a colonoscopy within 2 weeks of Visit 1 or are scheduled to have a colonoscopy during their participation in the study.
14. Subjects who withdraw consent at any time prior to completion of Visit 1 procedures

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2016-06; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, Study Director — Braintree Laboratories, Inc.
Locations (73):
- United States (73):
  - Braintree Research Site 43, Birmingham, Alabama
  - Braintree Research Site 30, Peoria, Arizona
  - Braintree Research Site 40, Phoenix, Arizona
  - Braintree Research Site 52, Phoenix, Arizona
  - Braintree Research Site 26, Phoenix, Arizona
  - Braintree Research Site 56, Fayetteville, Arkansas
  - Braintree Research Site 4, Little Rock, Arkansas
  - Braintree Research Site 51, Anaheim, California
  - Braintree Research Site 54, Fountain Valley, California
  - Braintree Research Site 8, Fresno, California
  - Braintree Research Site 71, Long Beach, California
  - Braintree Research Site 74, Oceanside, California
  - Braintree Research Site 59, Sacramento, California
  - Braintree Research Site 28, Sacramento, California
  - Braintree Research Site 68, Brooksville, Florida
  - Braintree Research Site 36, Fort Myers, Florida
  - Braintree Research Site 22, Homestead, Florida
  - Braintree Research Site 5, Jacksonville, Florida
  - Braintree Research Site 23, Jacksonville, Florida
  - Braintree Research Site 63, Miami, Florida
  - Braintree Research Site 29, Orlando, Florida
  - Braintree Research Site 65, Orlando, Florida
  - Braintree Research Site 13, Ormond Beach, Florida
  - Braintree Research Site 20, St. Petersburg, Florida
  - Braintree Research Site 39, St. Petersburg, Florida
  - Braintree Research Site 31, Tampa, Florida
  - Braintree Research Site 41, West Palm Beach, Florida
  - Braintree Research Site 57, Blue Ridge, Georgia
  - Braintree Research Site 48, Boise, Idaho
  - Braintree Research Site 50, Evansville, Indiana
  - Braintree Research Site 55, Lafayette, Indiana
  - Braintree Research Site 38, Wichita, Kansas
  - Braintree Research Site 64, Edgewood, Kentucky
  - Braintree Research Site 73, Lake Charles, Louisiana
  - Braintree Research Site 49, St Louis, Missouri
  - Braintree Research Site 19, Omaha, Nebraska
  - Braintree Research Site 21, Omaha, Nebraska
  - Braintree Research Site 69, Henderson, Nevada
  - Braintree Research Site 1, Las Vegas, Nevada
  - Braintree Research Site 44, Las Vegas, Nevada
  - Braintree Research Site 34, Las Vegas, Nevada
  - Braintree Research Site 7, Belvidere, New Jersey
  - Braintree Research Site 53, Trenton, New Jersey
  - Braintree Research Site 10, Albuquerque, New Mexico
  - Braintree Research Site 27, Brooklyn, New York
  - Braintree Research Site 25, Great Neck, New York
  - Braintree Research Site 61, Williamsville, New York
  - Braintree Research Site 45, Greensboro, North Carolina
  - Braintree Research Site 47, Winston-Salem, North Carolina
  - Braintree Research Site 2, Beavercreek, Ohio
  - Braintree Research Site 76, Cincinnati, Ohio
  - Braintree Research Site 3, Columbus, Ohio
  - Braintree Research Site 60, Columbus, Ohio
  - Braintree Research Site 14, Huber Heights, Ohio
  - Braintree Research Site 46, Oklahoma City, Oklahoma
  - Braintree Research Site 16, Oklahoma City, Oklahoma
  - Braintree Research Site 18, Lansdale, Pennsylvania
  - Braintree Research Site 75, Charleston, South Carolina
  - Braintree Research Site 17, Greer, South Carolina
  - Braintree Research Site 42, Myrtle Beach, South Carolina
  - Braintree Research Site 24, Spartanburg, South Carolina
  - Braintree Research Site 72, Spartanburg, South Carolina
  - Braintree Research Site 9, Summerville, South Carolina
  - Braintree Research Site 37, Chattanooga, Tennessee
  - Braintree Research Site 67, Tullahoma, Tennessee
  - Braintree Research Site 11, Austin, Texas
  - Braintree Research Site 33, Carrollton, Texas
  - Braintree Research Site 62, Channelview, Texas
  - Braintree Research Site 70, Houston, Texas
  - Braintree Research Site 35, Salt Lake City, Utah
  - Braintree Research Site 12, St. George, Utah
  - Braintree Research Site 66, West Jordan, Utah
  - Braintree Research Site 6, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BLI801 Laxative (High Dose) | BLI801 Laxative (Mid Dose) | BLI801 Laxative (Low Dose) | BLI801 Placebo
Started | 114 | 105 | 115 | 100
Completed | 101 | 90 | 100 | 90
Not Completed | 13 | 15 | 15 | 10

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population is based on the modified Intent-to-Treat population which includes patients who were randomized and took at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | BLI801 Laxative (High Dose) | BLI801 Laxative (Mid Dose) | BLI801 Laxative (Low Dose) | BLI801 Placebo | Total
Number analyzed (Participants) | 114 | 104 | 114 | 99 | 431
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (9.03) | 53.8 (10.43) | 53.4 (10.62) | 55.7 (10.61) | 54.6 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 69 | 80 | 71 | 289
  Male | 45 | 35 | 34 | 28 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 10 | 4 | 33
  Not Hispanic or Latino | 104 | 95 | 104 | 95 | 398
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: % of Subjects With Treatment Response
Description: Treatment response is defined as subjects who are weekly responders for at least 9 out of 12 weeks, with at least 3 of these weeks occurring in the last 4 weeks of treatment. A weekly responder is a subject who has ≥ 3 spontaneous bowel movements (SBMs) and an increase from baseline of > 1 SBM in that week.
Time Frame: 12 weeks
Population: The Primary Efficacy Analysis Population is based on the modified Intent-to-Treat population which includes patients who were randomized and took at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | BLI801 Laxative (High Dose) | BLI801 Laxative (Mid Dose) | BLI801 Laxative (Low Dose) | BLI801 Placebo
Number analyzed (Participants) | 114 | 104 | 114 | 99
Participants
  Success | 42 | 34 | 30 | 20
  Fail | 72 | 70 | 84 | 79
Statistical Analysis 1: Comparison: BLI801 Laxative (High Dose) vs BLI801 Laxative (Mid Dose) vs BLI801 Laxative (Low Dose) vs BLI801 Placebo; Test type: Superiority; p = 0.034, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 98 days
Description: The Adverse Event Population is based on the modified Intent-to-Treat population which includes patients who were randomized and took at least 1 dose of study medication.
Arm/Group | BLI801 Laxative (High Dose) | BLI801 Laxative (Mid Dose) | BLI801 Laxative (Low Dose) | BLI801 Placebo
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/104 | 0/114 | 0/99
Serious Adverse Events (participants affected / at risk) | 3/114 | 2/104 | 3/114 | 2/99
Other Adverse Events (participants affected / at risk) | 24/114 | 15/104 | 23/114 | 20/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLI801 Laxative (High Dose) (N=114) | BLI801 Laxative (Mid Dose) (N=104) | BLI801 Laxative (Low Dose) (N=114) | BLI801 Placebo (N=99)
Alcohol abuse secondary to worsening of depression and worsening of anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Worsening of syncope (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Worsening of atrial fibrilation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Takotsubo cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Opioid withdrawal (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atypical chest pain of musculoskeletal origin (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Worsening of chronic back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Worsening of cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain substernal pressure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Exacerbation vertigo (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
High ALT Values (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
High AST Values (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLI801 Laxative (High Dose) (N=114) | BLI801 Laxative (Mid Dose) (N=104) | BLI801 Laxative (Low Dose) (N=114) | BLI801 Placebo (N=99)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 1 (1) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 3 (3) | 5 (5) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 3 (3) | 6 (6) | 5 (5)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 6 (6) | 3 (3) | 6 (6) | 5 (5)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT02822508/Prot_SAP_000.pdf